CLINICAL TRIAL: NCT02354456
Title: An Epidemiological Study to Evaluate the Use of Vitamin K Antagonists and New Oral Anticoagulants Among Nonvalvular Atrial Fibrillation Patients in Turkey
Brief Title: Atrial Fibrillation in Turkey: Epidemiologic Registry-2
Acronym: AFTER-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hasan Kaya, Associate Professor of Cardiology, Dicle University
Other Study IDs: DicleU
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; epidemiology; antiocaogulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial fibrillation (AF) is one of the most common cause of preventable ischemic stroke and associated with increased cardiovascular morbidity and mortality. Our previous AFTER study demonstrated the general epidemiological data about the patients with valvular and nonvalvular AF in Turkey. However, data is lacking about the use of new oral anticoagulants (NOACs), time in therapeutic INR range (TTR) in vitamin K antagonist users and AF management modality in our country. In this multicenter trial the investigators aimed to analyze, follow and evaluate the epidemiological data in non-valvular AF patients.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cause of preventable stroke and strongly associated with increased cardiovascular morbidity and mortality with a prevalence of 1-2% in general population.The first multicenter trial in AF patients in our country, Atrial Fibrillation in Turkey: Epidemiologic Registry (AFTER) study, showed that 40% of non-valvular AF patients were on warfarin therapy with an effective INR rate of 37% and the most frequent cause of warfarin underuse was physician neglect. Yet, the use of new oral anticoagulants, time in therapeutic INR range (TTR) in warfarin users and the main management modality (rhythm or rate control) in AF patients have not been studied in Turkey. Therefore, in this multicenter trial, we aimed to assess the extent of effective anticoagulant use (by means of TTR) and epidemiological characteristics of the nonvalvular AF patients with the use of new oral anticoagulants (NOACs) in clinical practice in addition to increased awareness provided by AFTER study.

AFTER-2 study is planned as a prospective, observational and multicenter study with a 6 month and 1-year follow-up of the patients. A total of 4100 patients in 42 centers reflecting the population of the twelve regions of our country according to the Nomenclature of Territorial Units for Statistics will be included in the study.

The detailed characteristics of the patients with non-valvular AF, the rates and kind of oral anticoagulant use, the effect of increased awareness and NOACs on anticoagulant use rate, TTR in warfarin using patients and the bleeding risks of the patients will be determined in this study. At the end of the study, we will question the patients in terms of major adverse events and analyze the independent predictors of these events.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult non-valvular AF patients applied to the cardiology clinics with at least one attack of AF identified on electrocardiography without rheumatic mitral valve stenosis and prosthetic valve disease

Exclusion Criteria:

* Patients who will refuse to be a participant or will not sign the consent form

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nonvalvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Number of dead patients | 1 year
Number of patients with stroke | 1 year
Number of patients with major haemorrhage | 1 year
Number of hospitalization | 1 year

SECONDARY OUTCOMES:
Number of patients with time in therapeutic INR range | 1 year
  Time in therapeutic INR range calculated according to Rosendaal method

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Ertas, Assoc. Prof., Principal Investigator — Dicle University School of Medicine
Locations (1):
- Dicle Üniversity School of Medicine, Diyarbakır, Turkey (Türkiye)

REFERENCES:
- [Background] Kaya H, Ertas F, Kaya Z, Kahya Eren N, Yuksel M, Koroglu B, Kose N, Yildiz A, Cimen T, Ulgen MS. Epidemiology, anticoagulant treatment and risk of thromboembolism in patients with valvular atrial fibrillation: Results from Atrial Fibrillation in Turkey: Epidemiologic Registry (AFTER). Cardiol J. 2014;21(2):158-62. doi: 10.5603/CJ.a2013.0085. Epub 2013 Jun 25. PMID 23799558
- [Background] Ertas F, Eren NK, Kaya H, Aribas A, Acar G, Kanadasi M, Gedik S, Oylumlu M, Yuksel M, Ulgen MS; AFTER Investigators. The atrial fibrillation in Turkey: Epidemiologic Registry (AFTER). Cardiol J. 2013;20(4):447-52. doi: 10.5603/CJ.a2013.0055. Epub 2013 May 15. PMID 23677730
- [Background] Connolly SJ, Wallentin L, Ezekowitz MD, Eikelboom J, Oldgren J, Reilly PA, Brueckmann M, Pogue J, Alings M, Amerena JV, Avezum A, Baumgartner I, Budaj AJ, Chen JH, Dans AL, Darius H, Di Pasquale G, Ferreira J, Flaker GC, Flather MD, Franzosi MG, Golitsyn SP, Halon DA, Heidbuchel H, Hohnloser SH, Huber K, Jansky P, Kamensky G, Keltai M, Kim SS, Lau CP, Le Heuzey JY, Lewis BS, Liu L, Nanas J, Omar R, Pais P, Pedersen KE, Piegas LS, Raev D, Smith PJ, Talajic M, Tan RS, Tanomsup S, Toivonen L, Vinereanu D, Xavier D, Zhu J, Wang SQ, Duffy CO, Themeles E, Yusuf S. The Long-Term Multicenter Observational Study of Dabigatran Treatment in Patients With Atrial Fibrillation (RELY-ABLE) Study. Circulation. 2013 Jul 16;128(3):237-43. doi: 10.1161/CIRCULATIONAHA.112.001139. Epub 2013 Jun 14. PMID 23770747
- [Background] Yamashita T, Inoue H, Okumura K, Atarashi H, Origasa H; J-RHYTHM Registry Investigators. Warfarin anticoagulation intensity in Japanese nonvalvular atrial fibrillation patients: a J-RHYTHM Registry analysis. J Cardiol. 2015 Mar;65(3):175-7. doi: 10.1016/j.jjcc.2014.07.013. Epub 2014 Aug 26. PMID 25169015
- [Derived] Ertas F, Kaya H, Yildiz A, Davutoglu V, Kiris A, Dinc L, Kafes H, Avci A, Calapkorur B, Ertas G, Gul M, Kahraman Ay N, Bulur S, Durukan M, Eren M, Ilhan I, Kucuk M, Ozpelit E, Simsek H, Ucar FM, Yildiz A, Sahin DY, Ayhan E, Caglayan CE, Gungor H, Ozyurtlu F, Sen N, Vatan B, Vatansever F, Kobat MA, Temiz A, Taylan G, Donmez I, Erkus ME, Soylemez S, Zengin H, Gunduz M, Tuncez A, Karavelioglu Y, Gokdeniz T, Koza Y, Aktop Z, Katlandur H, Karaca Ozer P, Yuksel M, Acet H, Cil H, Alan S, Toprak N. An epidemiological study to evaluate the use of vitamin K antagonists and new oral anticoagulants among non-valvular atrial fibrillation patients in Turkey- AFTER-2 study design. Turk Kardiyol Dern Ars. 2015 Mar;43(2):169-77. doi: 10.5543/tkda.2015.35984. PMID 25782122